CLINICAL TRIAL: NCT02241460
Title: A Double-Blind, Placebo-Controlled, Randomized Study to Evaluate the Efficacy of Promescent Lidocaine Spray in Men With Premature Ejaculation
Brief Title: Efficacy of Promescent Lidocaine Spray in Men With Premature Ejaculation
Acronym: Promescent
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eugene Y Rhee, MD (Other)
Responsible Party: Sponsor-Investigator, Eugene Y Rhee, MD, Chief, Department of Urologic Surgery, Kaiser Permanente
Organization: Kaiser Permanente (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Promescent; KPSC IRB 6428 (Other: Kaiser Permanente Southern California Institutional Review Board)
Record Dates: First submitted 2014-05-12; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Premature Ejaculation
Keywords: Premature Ejaculation; Lidocaine
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Promescent Lidocaine Spray (Active Comparator): Double-Blind Treatment Period: 3 cycles (3 weeks each); 1 week wash-out between each cycle Open-Label Treatment Period: 4 cycles (1 week each); no wash-out
  Interventions: Drug: Promescent Lidocaine Spray
- Placebo (Placebo Comparator): Double-Blind Treatment Period: 3 cycles (3 weeks each); 1 week wash-out between each cycle Open-Label Treatment Period: 4 cycles (1 week each); no wash-out
  Interventions: Drug: Placebo; Drug: Promescent Lidocaine Spray

INTERVENTIONS:
Drug: Placebo — During the Double-Blind Treatment Period, patients randomized to placebo will receive three cycles of Promescent. The first and second cycle consists of three weeks of treatment using 30 mg and 50 mg, followed by one week of washout. The third cycle consists of three weeks of treatment using 70 mg. During the Open-Label Treatment Period, the patient will receive four weeks of Promescent (active treatment) in one-week cycles: 30 mg, 50 mg, 70 mg, and patient's self-selected dose.
  Arms: Placebo
Drug: Promescent Lidocaine Spray — During the Double-Blind Treatment Period, patients randomized to active treatment will receive three cycles of Promescent. The first and second cycle consists of three weeks of treatment using 30 mg and 50 mg, followed by one week of washout. The third cycle consists of three weeks of treatment using 70 mg, followed by four weeks of treatment during the Open-Label Treatment Period using patient's self-selected dose.

SUMMARY:
The purpose of this study is to evaluate the efficacy of treatment with Promescent Lidocaine Spray compared with placebo in patients with premature ejaculation.

DETAILED DESCRIPTION:
Promescent Lidocaine Spray is a non-prescription drug that is marketed under an over-the-counter drug monograph (21 CFR Section 348.10 Subpart B (a)(2)) for male genital desensitizing drug products. In addition the evaluating the efficacy of treatment with Promescent, this study will evaluate patients' subjective distress, perception of improvement and optimal dose, and safety and tolerability of Promescent for patients with premature ejaculation and their respective partners.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent before screening.
* Subject is a male, 18 years of age or older.
* Subject meets the diagnostic criteria for premature ejaculation as defined by the DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision; 2000).
* Subject has a stable, monogamous, heterosexual relationship and sexually active for at least the last 6 months.
* Subject and partner are willing and able to engage in sexual intercourse.

Exclusion Criteria:

* Subject has never achieved an intravaginal ejaculation during the past 6 months (i.e., always ejaculates prior to penetration).
* Subject has other forms of ejaculatory dysfunction (e.g., retrograde ejaculation, anejaculation, painful ejaculation).
* In the opinion of the investigator, the subject has a condition or is in a situation that may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's ability to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Intravaginal Ejaculatory Latency Time (IELT) in seconds | Week 11
  The primary efficacy outcome is the proportion of subjects that achieve a mean IELT of greater than 90 seconds at Week 3, 7, and 11.

SECONDARY OUTCOMES:
Subjective distress | Week 3, 7, and 11
Perception of improvement in premature ejaculation | Week 3, 7, and 11
Perceived optimal dosage of treatment | Week 3, 7, and 11
Adverse events/reactions to treatments | Week 11

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Y Rhee, MD, MBA, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente, Los Angeles, California
  - Kaiser Permanente, San Diego, California